CLINICAL TRIAL: NCT05757622
Title: Electroencephalogram Based Real-Time Sedation Level Prediction Using Artificial Intelligence
Brief Title: Electroencephalogram Based Real-Time Sedation Level Prediction
Acronym: EBSPA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 16097
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Procedural Sedation
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Propofol — Procedural sedation provided with propofol and remifentanil using target controlled infusions
Drug: Remifentanil — Procedural sedation provided with propofol and remifentanil using target controlled infusions

SUMMARY:
This is an observational pilot study. Patients undergoing elective surgery or Cath lab interventions under general anesthesia or procedural sedation at the department of anesthesiology at the UMCG will be enrolled.

1. Recruitment procedure:

   Patients identified as eligible for the study by research/clinical staff will be enrolled after written informed consent. Clinical staff involved in this study will approach the patient for obtaining informed consent prior to the scheduled procedure, according to the UMCG´s daily published OR/Cath lab schedule. Patients enrolled in this study will receive standard clinical care, as defined in the standard operating procedures of the department of Anesthesiology.
2. Monitor and recording set up:

   1. A vital sign monitor will continuously record routine physiological data, including ECG, noninvasive and/or invasive blood pressure (blood pressure cuff and/or arterial line), and pulse oximetry.
   2. The noninvasive EEG-monitor A disposable sensor will be attached to the forehead of the patient and passive recording of EEG and physiological data will begin prior to induction of anesthesia at the OR or Cath lab.
   3. Vital sign monitor and EEG-monitor used for this study are mounted permanently on the anesthesia machine and sedation workstation which is used routinely at the department of Anesthesiology and data obtained are directly streamed to the UMCG patient data record system , and stored monitor for case-based wave analysis.
3. Sedation/Pain assessments:

As per routine clinical practice, the investigators will use Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S) scoring system for sedation assessment system for pain assessment. During each assessment MOAA/S scores will be determined prior to induction of anesthesia or sedation, during the procedure, and after the procedure until the patient leaves the operating room/cath lab.

DETAILED DESCRIPTION:
This is an observational pilot study. Patients undergoing elective surgery or Cath lab interventions under general anesthesia or procedural sedation at the department of anesthesiology at the UMCG will be enrolled.

1. Recruitment procedure:

   Patients identified as eligible for the study by research/clinical staff will be enrolled after written informed consent. Clinical staff involved in this study will approach the patient for obtaining informed consent prior to the scheduled procedure, according to the UMCG´s daily published OR/Cath lab schedule. Patients enrolled in this study will receive standard clinical care, as defined in the standard operating procedures of the department of Anesthesiology.
2. Monitor and recording set up:

   1. A vital sign monitor will continuously record routine physiological data, including ECG, noninvasive and/or invasive blood pressure (blood pressure cuff and/or arterial line), and pulse oximetry.
   2. The noninvasive EEG-monitor A disposable sensor will be attached to the forehead of the patient and passive recording of EEG and physiological data will begin prior to induction of anesthesia at the OR or Cath lab.
   3. Vital sign monitor and EEG-monitor used for this study are mounted permanently on the anesthesia machine and sedation workstation which is used routinely at the department of Anesthesiology and data obtained are directly streamed to the UMCG patient data record system , and stored in the monitor for case-based wave analysis.
3. Sedation/Pain assessments:

As per routine clinical practice, the investigators will use Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S) scoring system for sedation assessment at each level of sedation. During each assessment , MOAA/S scores will be determined prior to induction of anesthesia or sedation, during the procedure, and after the procedure until the patient leaves the operating room/cath lab.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, undergoing elective procedures under general anesthesia or procedural sedation

Exclusion Criteria:

* Deemed unsuitable for selection by the research team or service care providers due to any medical, legal, social, or interpersonal issues that would either compromise the study or the routine care of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years, undergoing elective procedures under general anesthesia or procedural sedation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
EEG | From 5 minutes prior to start if induction to full awakening
  EEG recordings during procedural sedation
Vital signs | From 5 minutes prior to start if induction to full awakening
  Changes in Vital signs associated with the level of procedural sedation
MOAAS score | From 5 minutes prior to start if induction to full awakening
  sedation depth scoring using the MOAAS score

IPD SHARING:
Plan to Share IPD: Undecided